CLINICAL TRIAL: NCT04651023
Title: Shanghai Meiji Health Science and Technology Co., Ltd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Meiji Health Science and Technology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zai-Si Ji, phD, Principal Investigator, Shanghai Meiji Health Science and Technology Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ShanghaiMHST
Record Dates: First submitted 2020-11-16; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Over Weight People

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): During the 12-week study period, the participants consumed two bottles (2 *200 mL) of the experimental beverage (0g NnEx) per day with or after meals.
  Interventions: Dietary Supplement: Nelumbo nucifera Leaf Extract
- low concentration of NnEx group (Experimental): During the 12-week study period, the participants consumed two bottles (2 *200 mL) of the experimental beverage (1g NnEx) per day with or after meals.
  Interventions: Dietary Supplement: Nelumbo nucifera Leaf Extract
- high concentration of NnEx group (Experimental): During the 12-week study period, the participants consumed two bottles (2 *200 mL) of the experimental beverage (2g NnEx) per day with or after meals.
  Interventions: Dietary Supplement: Nelumbo nucifera Leaf Extract

INTERVENTIONS:
Dietary Supplement: Nelumbo nucifera Leaf Extract — Hot water extracted Nelumbo nucifera Leaf, mainly containing quercetin and quercetin 3-O-glucuronide.

SUMMARY:
Investigators performed a randomized double-blind trial to determine the effects of long-term NnEx ingestion in patients with overweight or obesity. Ninety-five participants (23<BMI<30 kg/m2) were randomly allocated to three groups: a control group, a 1 g/day NnEx group, and a 2 g/day NnEx group. The effects of the consumption of 2 g/day or 1 g/day NnEx for 12 weeks on indices of adiposity and fasting blood metabolic parameters were compared with those of no consumption of NnEx.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) of 23-30 kg/m2
* Has no history of using any antidiabetic medication
* Absence of liver, kidney, or heart disease
* Absence of food allergy and daily tea consumption <2 L
* Meet all of the above criteria and to follow the instructions given during the study.

Exclusion Criteria:

* Testing delayed for >1 week without justification
* Difficulty attending the hospital on the required days
* Lack of data regarding the times of beverage consumption for over 5% of the study
* Abnormal overeating
* Test results believed to be unreliable because of the lack of provision of diet and exercise reports during the fasting period
* Difficulty drawing blood
* Poor confidence in the test data

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2009-01-10 (Actual); Primary Completion 2009-05-15 (Actual); Study Completion 2009-06-20 (Actual)

PRIMARY OUTCOMES:
Changes in anthropometrix indices during the study | baseline, 6 weeks, 12 weeks
  weight in kilograms
Changes in anthropometrix indices during the study | baseline, 6 weeks, 12 weeks
  height in meters
Changes in anthropometrix indices during the study | baseline, 6 weeks, 12 weeks
  body fat in percentage
Changes in anthropometrix indices during the study | baseline, 6 weeks, 12 weeks
  visceral fat in percentage
Changes in anthropometrix indices during the study | baseline, 6 weeks, 12 weeks
  waist in centimeters
Changes in anthropometrix indices during the study | baseline, 6 weeks, 12 weeks
  hip in centimeters

SECONDARY OUTCOMES:
Changes in fasting biochemical indices during the study | baseline, 6 weeks, 12 weeks
  glucose in mmol/L
Changes in fasting biochemical indices during the study | baseline, 6 weeks, 12 weeks
  HbA1c in mmol/L
Changes in fasting biochemical indices during the study | baseline, 6 weeks, 12 weeks
  TG in mmol/L
Changes in fasting biochemical indices during the study | baseline, 6 weeks, 12 weeks
  FFA in mmol/L
Changes in fasting biochemical indices during the study | baseline, 6 weeks, 12 weeks
  T-cho in mmol/L
Changes in fasting biochemical indices during the study | baseline, 6 weeks, 12 weeks
  HDL-cho in mmol/L
Changes in fasting biochemical indices during the study | baseline, 6 weeks, 12 weeks
  LDL-cho in mmol/L
Changes in fasting biochemical indices during the study | baseline, 6 weeks, 12 weeks
  ASP in mmol/L
Changes in fasting biochemical indices during the study | baseline, 6 weeks, 12 weeks
  BUN in mmol/L